CLINICAL TRIAL: NCT03566342
Title: Optimal Regimen of Patient-controlled Epidural Analgesia in Laboring Patients Receiving Combined Spinal and Epidural Analgesia (CSE)
Brief Title: Optimal Regimen of Patient-controlled Epidural Analgesia in Laboring Patients
Acronym: PCEA
Status: Terminated | Type: Observational
Why Stopped: Preliminary analysis of data showed no significant findings
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, kalpana tyagaraj, Residency Program Director, Maimonides Medical Center
Other Study IDs: IRB #08/08/VA07
Record Dates: First submitted 2018-04-06; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: LABOR PAIN
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days

GROUPS / COHORTS (5):
- GROUP A: The PCEA solution will contain 0.1% Bupivacaine + 2.85 mcg/cc of Fentanyl. Basal infusion 7 ml/hour Demand dose 8ml Lockout ( number of doses per hour) 2 Lock out interval 30 minutes
- GROUP B: The PCEA solution will contain 0.1% Bupivacaine + 2.85 mcg/cc of Fentanyl. Basal infusion 7 ml/hour Demand dose 5ml Lockout ( number of doses per hour) 4 Lock out interval 15 minutes
- GROUP C: The PCEA solution will contain 0.1% Bupivacaine + 2.85 mcg/cc of Fentanyl. Basal infusion 7 ml/hour Demand dose 3ml Lockout ( number of doses per hour) 6 Lock out interval 10 minutes
- GROUP D: The PCEA solution will contain 0.1% Bupivacaine + 2.85 mcg/cc of Fentanyl. Basal infusion 14 ml/hour Demand dose 0 ml Lockout ( number of doses per hour) 0 Lock out interval 0 minutes
- GROUP E: The PCEA solution will contain 0.1% Bupivacaine + 2.85 mcg/cc of Fentanyl. Basal infusion 7 ml/hour Demand dose 7ml Lockout ( number of doses per hour) 3 Lock out interval 20 minutes

SUMMARY:
To test the efficacy of different recipes of epidural infusions used for providing pain relief during labor in parturients.

DETAILED DESCRIPTION:
In this prospective trial, the investigators would like to examine the efficacy of several different PCEA protocols in 250 parturients who receive CSE for labor pain. Any patient with failed epidural, delivery within 2 hours of epidural insertion, or Cesarean section will be excluded from the study. Each patient will be assigned to one of five groups (A - E), depending on the day of admission for delivery, excluding Friday and Saturday (observed religious holidays). Each group will have 50 patients.

ELIGIBILITY:
Inclusion Criteria:

Parturients receiving Combined Spinal epidural analgesia for labor pain relief.

Exclusion Criteria:

Any patient with failed epidural, delivery within 2 hours of epidural insertion, or Cesarean section will be excluded from the study.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — pregnant females
Study Population: Laboring women receiving combined spinal epidural analgesia for pain relief
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2007-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Pain scores | 24 to 48 hours.
  From each patient investigators will collect pain scores to assess the severity of labor pain, using the Visual Analog Scale (VAS) scale, 1-10. VAS score of 1 is considered minimal pain and VAS score of 10 is considered as the maximum pain.

SECONDARY OUTCOMES:
Number of boluses | 24 to 48 hours
  From each patient the investigators will obtain information on total number of boluses of the epidural medication used
Amount of medication used | 24 to 48 hours
  From each patient the investigators will obtain information regarding the total amount of medications used in mls from reviewing the history on the PCEA pump.
Motor block | 24 to 48 hours.
  For each patient, the investigators will obtain information regarding degree of motor block using the Modified Bromage scale.
  Modified Bromage score:
  1. Complete block (unable to move feet or knees)
  2. Almost complete block (able to move feet only)
  3. Partial block (just able to move knees)
  4. Detectable weakness of hip flexion while supine (full flexion of knees)
  5. No detectable weakness of hip flexion while supine
  6. Able to perform partial knee bend
Height of the patient | At recruitment of the patient in to the study
  From each patient the investigators will obtain information on height in inches.
Weight of the patient | At recruitment of the patient in to the study
  From each patient the investigators will obtain information on weight in pounds
Overall patient satisfaction | 24 to 48 hours
  From each patient investigators will collect satisfaction scores to assess degree of satisfaction, using the Visual Analog Scale (VAS) scale, 1-10. VAS score of 1 is considered minimal satisfaction and VAS score of 10 is considered as the maximum satisfaction.
Mode of delivery | 24 to 48 hours
  From each patient the investigators will obtain information regarding mode of delivery- vaginal delivery or C-Section

CONTACTS AND LOCATIONS:
Overall Officials: KALPANA TYAGARAJ, Principal Investigator — MAIMONIDES MEDICAL CENTER, 4802, 10TH AVENUE, BROOKLYN, NY-11219